CLINICAL TRIAL: NCT06235658
Title: Effects of Yoga on Physical and Psychological Outcomes in Older Patients Discharged From Cardiac Rehabilitation: A Pilot Study
Brief Title: Yoga in Older Cardiac Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Geunyeong Cha (Other)
Responsible Party: Sponsor-Investigator, Geunyeong Cha, Principal Investigator, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 86669
Record Dates: First submitted 2024-01-23; First posted 2024-02-01 (Actual); Last update posted 2024-03-26 (Actual); Status verified 2024-03

CONDITIONS: Cardiovascular Diseases in Old Age
Keywords: Physical Activity; Yoga; Mind-body therapies
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): Participants in the control group will not receive any intervention but will be provided with printed or electronic versions of the American Heart Association's 'Life's Essential 8' at baseline, which includes information on how to improve and maintain cardiovascular health.
- Online Yoga Intervention (Experimental): Participants in the intervention group will attend two virtual 60-minute gentle yoga sessions per week for 12 weeks.
  Interventions: Behavioral: Gentle Yoga

INTERVENTIONS:
Behavioral: Gentle Yoga — Participants will attend two virtual 60-minute gentle yoga sessions per week for 12 weeks. Each session will be conducted via videoconference using the Zoom platform, with participants joining from their homes.
  Arms: Online Yoga Intervention

SUMMARY:
The goal of this clinical trial is to compare, at 3 months, the effects of a yoga intervention on physical health, including balance, muscle strength, physical activity levels, cardiac autonomic function, and physical vulnerability, as well as psychological health, including depressive symptoms and anxiety, in cardiac patients who are older than 65 years old and randomized to the intervention or control group. The main questions aim to 1) determine if yoga can improve physical health outcomes such as balance, muscle strength, cardiac function, and physical vulnerability in older adults with cardiovascular disease, and 2) determine if yoga can positively impact psychological health, including reducing depressive symptoms and anxiety in this population. Participants in the intervention group will attend yoga sessions twice a week for three months. The intervention group will be asked to complete surveys and physical function assessments at the beginning and three months later. Researchers will compare the intervention group and the control group to see if there is any difference and improvement in physical and psychological health between the two groups.

ELIGIBILITY:
Inclusion Criteria:

* have a history of an acute myocardial infarction within the preceding year, stable angina, cardiac surgery (including heart transplantation, valve surgery, or coronary artery bypass), coronary artery angioplasty or stents, or heart failure (ejection fraction < 35%) diagnosed in the past year
* have completed facility-based cardiac rehabilitation program (phase CR-II) within 12 months
* can read and understand English
* have no major comorbidities limiting their ability to participate in a yoga intervention
* reside in Kentucky.

Exclusion Criteria:

* have incapacitating neurologic, orthopedic, or neoplastic conditions such as stroke paralysis, terminal cancer, or a cognitive disorder
* currently practice yoga
* have no home WIiFi access

Ages: 65 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-11-15 (Actual); Primary Completion 2024-12-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Recruitment rate | Three months
  The recruitment rate (%) will be calculated by dividing the total number of patients enrolled by approached eligible patients and then multiplying it by 100.
Retention rate | Three months
  The retention rate will be calculated by dividing the total number of patients by the number of patients who will complete the study and then multiplying it by 100.
Intervention adherence rate | Three months
  The intervention adherence rate will be calculated by dividing the total number of sessions attended by the total number of intervention sessions (i.e., 24) and multiplying that number by 100.
Intervention acceptability | Three months
  The investigators will use modified versions of the Treatment Acceptability Adherence Scale (TAAS) to assess acceptability of the yoga intervention at 3-months follow-up. The TAAS is a 10-item self-report questionnaire designed to evaluate treatment acceptability and adherence. Items are rated on a 7-point Likert-type scale (1 = disagree strongly; 7 = agree strongly). The total score is a sum of seven items, ranging from 10 to 49 where a higher score means greater adherence.
Intervention satisfaction | Three months
  The investigators will use modified versions of the Client Satisfaction Questionnaire (CSQ) to assess the satisfaction of the yoga intervention at 3-month follow-up. The CSQ is an 8-item self-report questionnaire to evaluate participant satisfaction with a specific intervention. Items are rated on a 4-point Likert-type scale (1 = very satisfied; 4= quite dissatisfied). The total score is the sum of eight items, ranging from 8 to 32, where a higher score indicates greater satisfaction with the intervention. This instrument was validated for patients and has internal consistency reliability.

SECONDARY OUTCOMES:
Change in Patient Health Questionnaire-9 | Baseline and Three months
  The Patient Health Questionnaire-9 (PHQ-9) was developed to correspond to symptoms used in the DSMV-IV to diagnose clinical depression. Nine symptoms are rated on a 4-point Likert scale (0 = 'Not at all; 3 = 'Nearly every day'), with possible total scores ranging from 0 to 27 and higher scores indicating higher levels of depressive symptoms.
Change in Brief Symptom Inventory | Baseline and Three months
  The Brief Symptom Inventory (BSI), anxiety index, consists of 6 items rated on a 5-point Likert scale (0 = not at all; 4 = extremely). The total score ranges from 0 to 24, with a higher score reflecting greater anxiousness.
Change in Vulnerable Elders Survey 13 | Baseline and Three months
  The Vulnerable Elders Survey 13 (VES-13) includes four dimensions: age, self-assessment of health, physical function, and living function. Each domain is scored differently. Age is scored as follows: 75-84 years = 1 point, ≥ 85 years = 3 points. Self-rated health is categorized into "fair and poor" or "good", "very good", or "excellent", with only the "fair and poor" category scoring 1 point. The total score ranges from 0 to 15, with higher scores indicating greater vulnerability.
Change in Short-term Heart Rate Variability | Baseline and Three months
  Short-term Heart Rate Variability (HRV) will be collected using the Polar H9 heart rate monitor (Polar Electro OY, Kempele, Finland). The investigator will send a reminder about the precautions to be taken (e.g., avoiding caffeine, alcohol, smoking, and intense physical activity, as these factors could affect the HRV measurement for successful HRV measurement the day before the scheduled test. The investigator will again ask if the instructions have been followed when they arrive for data collection.
  Study patients will be instructed to lay supine for 10 minutes without speaking and to remain as still as possible. The investigator will place the Polar H9 heart rate monitor on the center of the sternum to measure HRV. During HRV data collection, the study patients will also wear the ActiGraph on the waist because the Polar H9 communicates with the ActiGraph.
Change in Muscle strength | Baseline and Three months
  Muscle strengths will be measured using the handheld dynamometry (HHD, Lafayette dynamometer, model01165APP; Lafayette Instrument Company, Lafayette, Ind., USA). This device measures the peak force exerted in kilograms for five seconds during muscle contraction on hips, quadriceps, and biceps.
Change in Balance | Baseline and Three months
  Balance will be measured using an Inertial Measurement Unit device (DOTIMU; Xsens Technologies, Enschede., the Netherlands). The investigators attach the IMU sensor (a small device the size of a large watch face) to the participant's lower back at the level of L3 vertebra. Patients will be asked to take off their shoes and stand up on the mat with their hands on their hips for 30 seconds. The investigators will measure balance 3 times, with 30 seconds of rest between assessments. The total estimated time for the balance test is 3-5 minutes. All signal processing, subsequent feature extraction, and analysis will be performed using MATLAB version R2018B (The Mathworks Inc., Natick, MA, USA). The root-mean-square (RMS) value of the acceleration signal will be used to quantify the magnitude and trajectory of postural sway in each direction. The RMS of the magnitude vector of the 3-axis acceleration signal will be used as the summary score.
Change in Physical activity | Baseline and Three months
  Physical activity (PA) will be measured using actigraphy, the gold-standard for measuring physical activity. The investigator will use the ActiGraph (GT3X Link model), a triaxial instrument, which is the most widely used wearable accelerometer in clinical research. All patients will be instructed to wear the device for nine consecutive days, including at least one weekend day.

CONTACTS AND LOCATIONS:
Overall Officials: Debra K Moser, Ph.D, Study Chair — University of Kentucky
Locations (1):
- University of Kentucky, Lexington, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No